CLINICAL TRIAL: NCT06887283
Title: Essen Amyloidosis Registry
Acronym: EAR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: EAR-WDAZ1
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-03

CONDITIONS: Amyloidosis; Systemic; Amyloidosis Cardiac
Keywords: Amyloidosis; Transthyretin; Light chain amyloidosis; Neuropathy; Cardiomyopathy
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloid Neuropathies, Familial; Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Peripheral blood biobank samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Essen Amyloidosis Registry (EAR) is a prospective, observational registry designed to collect comprehensive clinical data on patients diagnosed with systemic amyloidosis. The registry aims to improve the understanding of disease progression, diagnostic pathways, and treatment outcomes. The registry is hosted at the University Hospital Essen and follows patients longitudinally. Inclusion is open to all patients with suspected or confirmed amyloidosis who provide informed consent.

DETAILED DESCRIPTION:
The Essen Amyloidosis Registry (EAR) is a single-center, prospective, observational registry designed to systematically collect clinical, laboratory, imaging, and outcome data from patients with suspected or confirmed systemic amyloidosis. The registry aims to improve the understanding of disease characteristics, diagnostic pathways, and treatment outcomes. While cardiac amyloidosis remains a main focus, EAR includes all forms of systemic amyloidosis, such as light-chain (AL) amyloidosis, transthyretin amyloidosis (ATTR, both hereditary and wild-type), and rarer subtypes.

Data collected include demographic information, medical history, comorbidities, diagnostic findings, treatment strategies, and longitudinal follow-up data on disease progression and therapy response. Standardized assessments include serial laboratory tests, cardiac and other imaging modalities (e.g., echocardiography, cardiac MRI, scintigraphy), and functional status evaluations. Routine quality-of-life assessments, as part of standard clinical practice, are also documented. Patients will not be required to complete additional study-specific questionnaires.

The registry further integrates a biobank component, in which biological samples are collected for biomarker analysis. Given the current limitations of available diagnostics-such as insufficient sensitivity for early disease detection and a lack of robust markers for therapy monitoring-these biospecimens may help identify new prognostic and predictive biomarkers.

EAR enables the analysis of risk factors, disease progression, and long-term outcomes based on real-world clinical data. The registry also serves as an internal quality control tool, ensuring standardized data collection and treatment monitoring. Patients remain under regular clinical follow-up, with routine evaluations every 3 to 6 months, depending on their disease stage and treatment regimen. These visits typically include resting ECGs, blood tests, imaging studies, and device checks (for patients with pacemakers or defibrillators).

The Essen Amyloidosis Registry aims to create a comprehensive dataset that can be utilized for future research projects. Sub-projects addressing specific scientific questions will be submitted as separate ethics applications. The study follows standard clinical care guidelines, with examinations performed according to established Standard Operating Procedures (SOPs) for amyloidosis management.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed amyloidosis (any)
* Written informed consent to participate in the study
* Age 18 years and above

Exclusion Criteria:

* Age < 18 years
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with suspected or confirmed amyloidosis treated at the University Hospital Duisburg-Essen are screened for inclusion. A particular focus of the registry lies on amyloid cardiomyopathy and amyloid polyneuropathy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall mortality or unplanned hospitalization for heart failure | 24 months
  Overall mortality or unplanned hospitalization for heart failure is defined as the primary endpoint. The time to the primary endpoint will be measured in days starting from the day of first diagnosis of cardiac amyloidosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The study is planned as a monocentric registry but is open to requests of scientific cooperation.